CLINICAL TRIAL: NCT02868021
Title: Blood Flow Restriction Exercise for Older Adults Undergoing Knee Replacement Surgery
Brief Title: Blood Flow Restriction Exercise Study
Acronym: BFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: University of Florida Clinical and Translational Science Institute (CTSI) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB201601042
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Osteoarthritis, Knee
Keywords: Elderly; Exercise
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Walking; Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NO-EX group (Placebo Comparator): Subjects allocated to the No Exercise (NO-EX) group will undergo: Strength testing, Short Physical Performance Battery (SPPB), Six-minute walk (SMW), Numerical pain scale, Self-assessed function and Six-minute walk (SMW) test. Intra-op muscle biopsies.
  Interventions: Device: Strength testing; Behavioral: Short Physical Performance Battery (SPPB); Behavioral: Six-minute walk (SMW); Behavioral: Numerical pain scale; Behavioral: Self-assessed function; Procedure: Muscle biopsies
- EX-BFR group (Experimental): Subjects allocated to the EX-BFR group will undergo baseline strength testing, Short Physical Performance Battery (SPPB), Numerical pain scale, Six-minute walk (SMW), Self-assessed function, and determination of 1 Repetition Maximum (1-RM). Blood flow restriction exercise, Borg Category Ratio 10 (Borg CR10) scale. Intra-op muscle biopsies.
  Interventions: Device: Strength testing; Behavioral: Short Physical Performance Battery (SPPB); Behavioral: Six-minute walk (SMW); Behavioral: Numerical pain scale; Behavioral: Self-assessed function; Procedure: Muscle biopsies; Device: Determination of 1 Repetition Maximum (1-RM); Device: Blood flow restriction exercise; Behavioral: Borg CR10 scale

INTERVENTIONS:
Device: Strength testing — Test the strength of subject's lower extremity muscles on the dynamometer system
Behavioral: Short Physical Performance Battery (SPPB) — The SPPB is a timed short distance walk, repeated chair stands, and balance test that measures lower extremity function.
Behavioral: Six-minute walk (SMW) — Subjects walk back and forth along a 100-ft hallway for six minutes after instructions to complete as many laps as possible.
Behavioral: Numerical pain scale — Measure pain using an 11-point numerical pain scale.
Behavioral: Self-assessed function — Using the Late Life Function and Disability Instrument.
Procedure: Muscle biopsies — During the course of the surgery two small muscle biopsies from the quadriceps muscle of the operative leg will be collected.
Device: Determination of 1 Repetition Maximum (1-RM) — Following the warm-up, subjects will attempt to complete one repetition of the leg press exercise at progressively greater resistance until a full repetition can no longer be performed. The weight of the last complete unassisted repetition will be recorded as the 1-RM.
  Arms: EX-BFR group
Device: Blood flow restriction exercise — Perform lower-extremity exercises (leg press, leg extension, leg curl, and calf extension) at an intensity of 30% of 1-RM with external compression applied to the proximal thigh of each leg.
  Arms: EX-BFR group
Behavioral: Borg CR10 scale — Following each exercise session, participants will provide a rating of perceived exertion (RPE) for the session according to the Borg CR10 scale.
  Arms: EX-BFR group

SUMMARY:
This pilot study will investigate the effects of blood flow restriction (BFR) exercise for up to 4-6 weeks prior to total knee arthroplasty (TKA) surgery in older patients to measure clinical outcomes such as strength, lower extremity function, and pain.

DETAILED DESCRIPTION:
The purpose of this study is to test the feasibility and efficacy of a low-resistance exercise protocol with blood flow restriction (BFR) using a tourniquet in the preoperative period of patients awaiting TKA. BFR exercise is a new exercise method that has not been studied in the perioperative period. The investigators will compare our intervention to a no-exercise group up to 4 - 6 weeks prior to surgery to determine if this type of exercise is feasible in the preoperative period and if BFR exercise will improve functional, physiological, and molecular outcomes when compared to patients without exercise.

ELIGIBILITY:
Inclusion Criteria:

* are scheduled for elective TKA for osteoarthritis
* are scheduled for unilateral joint replacement surgery only
* are able to give consent and follow instructions
* are willing to complete up to 15 study visits

Exclusion Criteria:

* patients below the age of 55 years old
* patients over the age of 80 years old
* patients who live in a radius greater than 45 miles from the University of Florida (a feasible distance to allow for transportation to and from the clinical center for assessment visits)
* patients with impaired cognitive function and mental disease, (e.g. diagnosis of Alzheimer's disease)
* patients with paraplegia/extremity amputation
* patients with end stage renal disease requiring dialysis
* patients with uncontrolled diabetes and insulin-dependent diabetes
* patients with uncontrolled cardiovascular disease e.g. (Classes of Heart Failure (CHF) New York Heart Association (NYHA) class 3 or higher, BP > 180/110 mmHg)
* patients with severe pulmonary disease requiring continuous oxygen therapy
* patients with active neoplasm
* patients with peripheral vascular disease or deep vein thrombosis (within the last 3 years)
* patients with structured exercise/Physical Therapy(PT)/Occupational Therapy (OT)/fitness program enrollment within 12 weeks prior to surgery and/or more than 2 hours per month on gym/fitness room exercises
* patients with BMI greater than 40 kg/m2
* patients with opioid use of more than 30 mg Morphine-equivalents per day
* patients with chronic oral steroid use
* patients with chronic anticoagulation (e.g. Plavix, Warfarin)
* patients with planned postoperative admission to a skilled nursing/inpatient rehab facility
* patients with ipsilateral joint disease involving hip, ankle or spine
* neurologic or other etiology of quadriceps wasting
* surgery within less than 4 weeks
* patients with comorbidities that the PI judges as not suitable for the study
* patients with a minimal mental status (MMSE) score below 24

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Changes between the two group assessed by muscle strength | Changes from baseline (pre-op) up to 2 weeks post-op
  Test the strength of subject's lower extremity muscles on the dynamometer system

SECONDARY OUTCOMES:
Changes between the two group assessed by Short Physical Performance Battery (SPPB) | Changes from baseline (pre-op) up to 2 weeks post-op
  SPPB is a validated test to measure lower extremity function a timed short distance walk, repeated chair stands, and balance test.
Changes between the two group assessed by Six-minute walk (SMW) test | Changes from baseline (pre-op) up to 2 weeks post-op
  SPPB is a validated test to measure lower extremity function a timed short distance walk, repeated chair stands, and balance test.
Changes between the two group assessed by pain | Changes from baseline (pre-op) up to 2 weeks post-op
  Measure pain using an 11-point numerical pain scale
Changes between the two group assessed by self-assessment outcomes | Changes from baseline (pre-op) up to 2 weeks post-op
  Assessed using the Late Life Function and Disability Instrument
Changes between the two group assessed by biological targets on the muscle tissue | Up to 4 hours (end of surgery)
  Analysis of the muscle tissue will focus on metabolism, inflammation, autophagy, apoptosis and other mechanisms of muscular atrophy.

CONTACTS AND LOCATIONS:
Overall Officials: Rene Przkora, MD, Principal Investigator — University of Florida
Locations (1):
- United States, Florida UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No